CLINICAL TRIAL: NCT05140746
Title: A Prospective Study on Predicting the Efficacy of Neoadjuvant Chemotherapy in Locally Advanced Gastric Cancer.
Brief Title: Prediction of Neoadjuvant Chemotherapy Efficacy in Locally Advanced Gastric Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PET-NAC-GC
Record Dates: First submitted 2021-11-08; First posted 2021-12-01 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET/CT for prediction of NAC efficacy (Experimental): 68Ga-FAPI-04 PET/CT and 18F-FDG PET/CT will be scanned before, during or after NAC.
  Interventions: Diagnostic Test: 68Ga-FAPI-04 PET/CT and 18F-FDG PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI-04 PET/CT and 18F-FDG PET/CT — Baseline 68Ga-FAPI-04 PET/CT and 18F-FDG PET/CT scans before NAC followed by abdomen 68Ga-FAPI-04 PET/CT and 18F-FDG PET/CT scans after one cycle of NAC treatment or before surgery.

SUMMARY:
This study intends to explore the value of 68Ga-FAPI-04 and 18F-FDG PET/CT in the evaluation of treatment response to neoadjuvant chemotherapy(NAC) for patients with locally advanced gastric cancer(LAGC).

DETAILED DESCRIPTION:
Before the start of NAC, baseline 68Ga-FAPI-04 PET/CT and 18F-FDG PET/CT scans will be scheduled in all enrolled patients. Next, the patients with resectable LAGC will receive NAC treatment, surgery will follow 3~6 weeks after finishing NAC. Abdomen 68Ga-FAPI-04 PET/CT and 18F-FDG PET/CT will be scheduled after one cycle of NAC treatment or before surgery. Imaging response measurements will be compared with the histopathological tumor regression grade (TRG) of the resection specimen as gold standard.

ELIGIBILITY:
Inclusion criteria

1. Age between 18-75 years.
2. Histologically confirmed gastric adenocarcinoma through gastroscopy.
3. Resectable gastric cancer.
4. ECOG performance status 0-1.
5. White blood count >4x109/L, Absolute neutrophil count (ANC) >2x109/L, Hemoglobin (Hb)>90g/L, Platelets >100x109/L.
6. Ejection Fraction>50%.
7. Serum bilirubin <1.5x ULN; ALT and AST <1.5x ULN.
8. Serum creatinine ≤1.5x ULN, or GFR> 60ml/min.
9. Agreement to participate in this study with informed consent form.
10. Willingness and ability to comply with the protocol for the duration of the study.
11. No children bearing petential in the next six months before enrollment.

Exclusion criteria

1. With second primary malignant diseases in past five years, exceptions include basal cell and squamous cell carcinoma of the skin that have been cured.
2. Known hypersensitivity reaction to chemotherapy drugs or with contraindications.
3. With severe disease or other unsuitable conditions determined by investigators. Inadequate organ function.
4. With uncontrollable diabetic or fasting blood glucose level ≥11 mmol/L on the test-day.
5. With severe mental symptoms, unconscious or unable to complete the examination.
6. Pregnancy or possibly pregnant woman, breastfeeding woman.
7. Lack of compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2024-09-10 (Estimated); Study Completion 2027-09-10 (Estimated)

PRIMARY OUTCOMES:
Prediction for NAC efficacy | Two weeks after surgery
  Predictive value of 68Ga-FAPI PET/CT and 18F-FDG PET/CT for LAGC in NAC response assessment.
Standardized uptake value(SUV) | Two weeks after surgery
  SUV of 68Ga-FAPI and 18F-FDG uptake on PET/CT images for primary gastric cancer.
Target-to-background ratio(TBR) | Two weeks after surgery
  68Ga-FAPI and 18F-FDG uptake ratio of primary gastric cancer to mediastinum blood pool on PET/CT images.

SECONDARY OUTCOMES:
Diagnostic efficacy for metastatic lymph nodes | Two weeks after surgery
  The sensitivity, specificity, NPV, PPV and accuracy of 68Ga-FAPI PET/CT for metastatic lymph nodes in comparison with those of 18F-FDG PET/CT.
Disease free survival | 5 years
  Disease free survival
Overall survival | 5 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Zhenggang Zhu, Principal Investigator — Ruijin Hospital
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Miao Y, Feng R, Yu T, Guo R, Zhang M, Wang Y, Hai W, Shangguan C, Zhu Z, Li B. Value of 68Ga-FAPI-04 and 18F-FDG PET/CT in Early Prediction of Pathologic Response to Neoadjuvant Chemotherapy in Locally Advanced Gastric Cancer. J Nucl Med. 2024 Feb 1;65(2):213-220. doi: 10.2967/jnumed.123.266403. PMID 38164574